CLINICAL TRIAL: NCT07251491
Title: Safety, Tolerability, Outcomes of Psilocybin for Depression (STOP Depression) in Veterans With Spinal Cord Injury
Brief Title: Psilocybin to Treat Depression in Spinal Cord Injury
Acronym: STOP
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Bronx Veterans Medical Research Foundation, Inc (Other); Usona Institute (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jill M. Wecht, Ed.D., Principal Investigator, James J. Peters Veterans Affairs Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 1872390; SC240097 (Other Grant/Funding Number: CDMRP Department of Defense)
Record Dates: First submitted 2025-09-30; First posted 2025-11-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injury; Depression - Major Depressive Disorder; Veteran
Keywords: Tetraplegia; Paraplegia; Psychosocial Wellbeing; Depression; Neuropathic Pain; Psychedelics
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia; Paraplegia; Depression; Neuralgia | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: psilocybin 5mg psilocybin 10mg psilocybin 25mg
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Psilocybin Low Dose (Experimental): Psilocybin 5mg
  Interventions: Drug: Psilocybin (Usona Institute)
- Psilocybin Medium Dose (Experimental): Psilocybin 10mg
  Interventions: Drug: Psilocybin (Usona Institute)
- Psilocybin High Dose (Experimental): Psilocybin 25mg
  Interventions: Drug: Psilocybin (Usona Institute)

INTERVENTIONS:
Drug: Psilocybin (Usona Institute) — Oral capsules
  Other Names: Magic Mushrooms

SUMMARY:
The main goal of this study is to determine if psilocybin is safe for use in people with SCI. The study will measure how people with SCI respond to three psilocybin doses: low (5mg), medium (10mg), and high (25mg).

The main question the study aims to answer is: does psilocybin increase the number and severity of adverse (bad) events reported by people with SCI? These may include pain, muscle spasms, symptoms of depression, and symptoms of low or high blood pressure. The investigators will also measure how well people with SCI tolerate the psychedelic experience, and compare responses between the low (5mg), medium (10mg), and high (25mg) doses.

Participants will:

* Agree to be enrolled in the study for up to 13 months.
* Agree to complete the seven (7) visits that are included in the psilocybin-assisted therapy.
* Agree to complete follow-up study visits, including in-person visits to the James J Peters VA Medical Center, located in the Bronx, New York and remote visits.
* Agree to keep a log of how they are feeling and any change in the frequency or severity of adverse events.

DETAILED DESCRIPTION:
Background: Depression may be explained partly by decreased signaling of serotonin in the nervous system. Psilocybin, the active component of 'magic mushrooms', is a drug that activates serotonin pathways in the nervous system. Some scientists think psilocybin could help people with major depression, but it is not currently approved as a medicine in the United States. People with spinal cord injuries (SCI) often feel depressed, even more commonly than people without injuries. People with SCI have not been included in psilocybin studies. The goals of this study are first to see if psilocybin can be safely administered, and to determine if psilocybin can help improve symptoms of depression in people with SCI. Study Goals: The investigators will look at how safe psilocybin is for people with SCI, how people with SCI respond to different doses, and whether it helps reduce the severity of depression and other problems, like pain or muscle spasms. The study team will also check to see if psilocybin improves quality of life and wellbeing. The study will track these effects for a year after participants receive psilocybin. Study Plan: Thirty people with chronic SCI with a depressive disorder will be asked to join-15 with paraplegia and 15 with tetraplegia. They will be split into three groups to try different psilocybin doses: low (5mg), medium (10mg), and high (25mg). The study will take a stepwise approach to safety, but participants will not know the dose of psilocybin they receive. There will be at least 16 study visits, including medical and mental health check-ups, psilocybin assisted therapy, primary study endpoint and follow-up visits. What Will Be Measured: The study focus is to see if psilocybin is safe and tolerable in people with SCI. The study will track side effects, how people feel, and any changes in mood, pain, medication use, or body reactions. Doctors will check for problems like chest pain, high blood pressure, and changes in suicidal thoughts. The study team will also measure satisfaction with the therapy, experiences during the psilocybin sessions, and changes in depression. Why It Matters: Some people wrongly believe depression is just a normal part of living with SCI, so their depression may not be adequately treated. Also, people with SCI often can't join trials of new treatments because they have other health problems. Psilocybin could help treat depression and may improve many body functions affected by SCI if it is shown to be safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent
* Spinal cord injury for at least 1 year
* Confirmed diagnosis of depression
* At least 22 years of age at time of consent
* At least 50 kg (110 lbs.) body weight
* Fully independent from ventilatory support (ventilator or diaphragm pacer)
* Fluent in speaking and reading English
* Able to swallow pills
* Agree to have study visits recorded with audio and video
* Agree to release outside medical and psychiatric records
* Able and willing to taper off antidepressant, under clinician supervision
* Agree to use adequate contraceptive methods

Exclusion Criteria:

* Are not able to give adequate informed consent
* Have used psilocybin or another psychedelic within 6 months
* Have received Electroconvulsive Therapy (ECT) within 12 weeks
* Have used ketamine within 12 weeks
* Have a history of Bipolar I Disorder
* Have a current eating disorder
* Have a current severe alcohol or cannabis use disorder within the 6 months
* Have an illicit drug or prescription drug substance use disorder within 12 months
* Current serious suicide risk
* History of heart attack, aneurysm, or stroke
* Uncontrolled hypertension
* Are pregnant or nursing

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by the Adverse Events Log. | Screening through study completion, an average of 13 months.
  The Adverse Events Log will be captured by the research team at screening, before and after medication taper (if needed), weekly during the taper, at each of the three preparatory and three integration sessions, at 44 days post dose, and at all remote and in-person follow-up visits; 16 assessments in total.

SECONDARY OUTCOMES:
Clinician rated change from baseline (V1) in the Montgomery-Asberg Depression Rating Scale (MADRS) score at 44(+/-7) days post psilocybin dose (V9). | Baseline to 44 days post psilocybin.
  The MADRS is a ten-item diagnostic questionnaire that includes questions related to symptoms of (1) apparent sadness; (2) reported sadness; (3) inner tension; (4) reduced sleep; (5) reduced appetite; (6) concentration difficulties; (7) lassitude; (8) inability to feel; (9) pessimistic thoughts; and (10) suicidal thoughts. Each item yields a score of 0 to 6, with higher scores reflecting more severe depression. MADRS scores correspond to 0-6 (normal or no depression), 7-19 (mild depression), 20-30 (moderate depression), 31-39 (severe depression), and 40-60 (extremely severe depression). Higher scores are indicative of higher levels of depression, range of scores 0-60.
Self reported change in depression severity score on the Beck Depression Inventory (BDI-II) from baseline (V1) to 44(+/-7) days post psilocybin (V9). | Baseline to 44 days post psilocybin.
  The BDI-II consists of four answer choices that are scored from 0 (no symptom) to 3 (severe symptom). Total BDI scores correspond to 0-9 (minimal depression), 10-18 (mild depression), 19-29 (moderate depression) and 30-63 (severe depression). Higher scores are indicative of higher levels of depression, range of scores 0-63.

OTHER OUTCOMES:
Change in self-reported levels of pain interference in daily life, overall mood, and sleep quality from baseline (V1) to 7 days post psilocybin (V7) using the International Spinal Cord Injury Pain Basic Data Set (iSCI-PBD). | Baseline to 7 days post psilocybin.
  The iSCI-PBD detects change in the number of painful condition types, the severity of pain, location of painful conditions, and pain interference in daily life, overall mood, and sleep quality. The outcome will include change in pain interference in daily life, overall mood, and sleep quality from baseline (V1) to 7 days post psilocybin (V7) using the iSCI-PBD with scores ranging from 0 (no interference) to 10 (extreme interference). Higher scores are indicative of higher levels of pain interference, range of scores 0-10.
Self-reported change in frequency and severity of spasms using the Penn Spasm Frequency Scale (PSFS) . | Baseline to 7 days post psilocybin.
  The PSFS is a self-report measure used to assess the perception (over a one-week time frame) of spasticity frequency on a 0 ("no spasm") to 4 ("spasms occurring more than 10 times per hour) scale, and severity on a 1 ("mild") to 3 ("severe") following SCI. The investigators will track change changes in spasms from baseline (V1) to 7 days post psilocybin (V7). Higher scores are indicative of higher levels of spasm frequency (score range 0-4) and spasm severity (score range 0-3).

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Wecht, EdD, Principal Investigator — James J Peters VA Medical Center
Locations (1):
- James J. Peters Department of Veterans Affairs Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
If data will not be shared it is due to restrictive policies within the VA.

REFERENCES:
- [Background] Lyes M, Yang KH, Castellanos J, Furnish T. Microdosing psilocybin for chronic pain: a case series. Pain. 2023 Apr 1;164(4):698-702. doi: 10.1097/j.pain.0000000000002778. Epub 2022 Sep 5. PMID 36066961
- [Background] Abrams SK, Rabinovitch BS, Zafar R, Aziz AS, Cherup NP, McMillan DW, Nielson JL, Lewis EC. Persons With Spinal Cord Injury Report Peripherally Dominant Serotonin-Like Syndrome After Use of Serotonergic Psychedelics. Neurotrauma Rep. 2023 Aug 22;4(1):543-550. doi: 10.1089/neur.2023.0022. eCollection 2023. PMID 37636336
- [Background] Liu Y, Collins C, Wang K, Xie X, Bie R. The prevalence and trend of depression among veterans in the United States. J Affect Disord. 2019 Feb 15;245:724-727. doi: 10.1016/j.jad.2018.11.031. Epub 2018 Nov 5. PMID 30699861
- [Background] Smith BM, Weaver FM, Ullrich PM. Prevalence of depression diagnoses and use of antidepressant medications by veterans with spinal cord injury. Am J Phys Med Rehabil. 2007 Aug;86(8):662-71. doi: 10.1097/PHM.0b013e318114cb6d. PMID 17667197
- [Background] Sloshower J, Skosnik PD, Safi-Aghdam H, Pathania S, Syed S, Pittman B, D'Souza DC. Psilocybin-assisted therapy for major depressive disorder: An exploratory placebo-controlled, fixed-order trial. J Psychopharmacol. 2023 Jul;37(7):698-706. doi: 10.1177/02698811231154852. Epub 2023 Mar 20. PMID 36938991
- [Background] Goodwin GM, Aaronson ST, Alvarez O, Atli M, Bennett JC, Croal M, DeBattista C, Dunlop BW, Feifel D, Hellerstein DJ, Husain MI, Kelly JR, Lennard-Jones MR, Licht RW, Marwood L, Mistry S, Palenicek T, Redjep O, Repantis D, Schoevers RA, Septimus B, Simmons HJ, Soares JC, Somers M, Stansfield SC, Stuart JR, Tadley HH, Thiara NK, Tsai J, Wahba M, Williams S, Winzer RI, Young AH, Young MB, Zisook S, Malievskaia E. Single-dose psilocybin for a treatment-resistant episode of major depression: Impact on patient-reported depression severity, anxiety, function, and quality of life. J Affect Disord. 2023 Apr 14;327:120-127. doi: 10.1016/j.jad.2023.01.108. Epub 2023 Feb 4. PMID 36740140
- [Background] Goodwin GM, Aaronson ST, Alvarez O, Arden PC, Baker A, Bennett JC, Bird C, Blom RE, Brennan C, Brusch D, Burke L, Campbell-Coker K, Carhart-Harris R, Cattell J, Daniel A, DeBattista C, Dunlop BW, Eisen K, Feifel D, Forbes M, Haumann HM, Hellerstein DJ, Hoppe AI, Husain MI, Jelen LA, Kamphuis J, Kawasaki J, Kelly JR, Key RE, Kishon R, Knatz Peck S, Knight G, Koolen MHB, Lean M, Licht RW, Maples-Keller JL, Mars J, Marwood L, McElhiney MC, Miller TL, Mirow A, Mistry S, Mletzko-Crowe T, Modlin LN, Nielsen RE, Nielson EM, Offerhaus SR, O'Keane V, Palenicek T, Printz D, Rademaker MC, van Reemst A, Reinholdt F, Repantis D, Rucker J, Rudow S, Ruffell S, Rush AJ, Schoevers RA, Seynaeve M, Shao S, Soares JC, Somers M, Stansfield SC, Sterling D, Strockis A, Tsai J, Visser L, Wahba M, Williams S, Young AH, Ywema P, Zisook S, Malievskaia E. Single-Dose Psilocybin for a Treatment-Resistant Episode of Major Depression. N Engl J Med. 2022 Nov 3;387(18):1637-1648. doi: 10.1056/NEJMoa2206443. PMID 36322843
- [Background] Khazaeipour Z, Taheri-Otaghsara SM, Naghdi M. Depression Following Spinal Cord Injury: Its Relationship to Demographic and Socioeconomic Indicators. Top Spinal Cord Inj Rehabil. 2015 Spring;21(2):149-55. doi: 10.1310/sci2102-149. Epub 2015 Apr 12. PMID 26364284
- [Background] Krause JS, Kemp B, Coker J. Depression after spinal cord injury: relation to gender, ethnicity, aging, and socioeconomic indicators. Arch Phys Med Rehabil. 2000 Aug;81(8):1099-109. doi: 10.1053/apmr.2000.7167. PMID 10943762